CLINICAL TRIAL: NCT05175911
Title: Implementation of the "Golden Hour", an Initial Standardized Stabilization of Preterm Less Than 31 Weeks and/or 1300 g : a Quality Improvement Study
Brief Title: Implementation of the Golden Hour for Preterm Infants : a Quality Improvement Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Liege (Other)
Responsible Party: Principal Investigator, Tribolet Sophie, Doctor, Centre Hospitalier Universitaire de Liege
Other Study IDs: Golden
Record Dates: First submitted 2021-12-01; First posted 2022-01-04 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Premature Birth
Keywords: premature birth; golden hour; 60 minutes
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- premature infants: premature infants less than 31 weeks of gestation or weighting less than 1300 g
  Interventions: Other: golden hour : an initial standardized stabilization

INTERVENTIONS:
Other: golden hour : an initial standardized stabilization — This is a quality improvement project to evaluate the implementation of "Golden hour", a standardized stabilization during the first hour of life in inborn preterm infants younger than 31 weeks of gestational age or weighting less than 1300 g in the NICU of the University of Liege.
  There is no comparative arm.

SUMMARY:
Effective initial stabilization of preterm neonates in the initial 60 minutes of life ("golden hour") was shown to improve outcomes. Keys components include anticipative and collaborative approach, respiratory support, thermal regulation and early initiation of parenteral nutrition. The objective is to complete the admission within 60 minutes of delivery.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants (< 31 weeks' gestation)
* Infants with expected weight less than 1300 g
* Inborn babies

Exclusion Criteria:

* Infants outborn
* Infants with major congenital anomalies (laparoschisis, omphalocèle, diaphragmatic hernia, …)
* Parental refusal

Max Age: 1 Hour | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature younger than 31 weeks of gestational age or less than 1300 g expected
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Completion of the procedure : closing time of the incubator | 1 hour
  Number of minutes of life at incubator closure
Glycemia at admission and within 24 hours | 24 hours
  blood glucose measurement on admission and then every 3 hours for the first 24 hours of life
Thermal stability : temperature at admission and at the end of the procedure | 1 hour
Mortality rate | 3 months

SECONDARY OUTCOMES:
Process of the procedure: | 1 hour
  Number of minutes of life at initiation of parenteral nutrition, caffeine and antibiotics administration.
Incidence of hypotension and bradycardia | 1 hour
Intubation rate and duration of mechanical ventilation | 3 months
  Number of hours of mechanical ventilation
Need for surfactant administration and time of administration | 3 days
  Number of hours of life at surfactant administration
Comorbidities of prematurity: NEC, BPD, ROP, sepsis, PDA, cPVL, IVH | 3 months
Duration of hospital stay (only if no transfer) | 3 months
Caregiver's perception of the procedure: stress… | 24 hours
  use of a questionnaire adapted from the "Teamwork Perceptions Questionnaire (T-TPQ)"
Parental experience of the procedure | 24 hours
Conditions of the procedure : realization during the night shift and team composition | 24 hours
  collection of the time and date of performance and the number of nurses, doctors, fellows,...

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No